CLINICAL TRIAL: NCT02945982
Title: A Randomized, Placebo-Controlled, Open-label, Multi-Center Study to Assess the Efficacy and Safety of Fuzheng Huayu Combined With Entecavir and Carvedilol in Moderate and Severe Cirrhotic Portal Hypertension Due to Hepatitis B Virus
Brief Title: Treatment of Moderate and Severe Cirrhotic Portal Hypertension Due to HBV With Fuzheng Huayu and Entecavir
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShuGuang Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other); Longhua Hospital (Other); Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Liu Chenghai, Professor, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGHLC20161023004
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Portal Hypertension
Keywords: Portal Hypertension; Fuzheng Huayu; Hepatitis B
MeSH Terms: conditions — Hypertension, Portal; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entecavir/Carvedilol (Placebo Comparator): Tablet with Entrcavir and Carvedilol
  Interventions: Drug: Entecavir+Carvedilol
- Entecavir/Carvedilol/ Fuzheng Huayu (Experimental): Tablet with Entrcavir and Carvedilol+ Tablet with Fuzheng Huayu
  Interventions: Drug: Entecavir+Carvedilol+ Fuzheng Huayu

INTERVENTIONS:
Drug: Entecavir+Carvedilol — The subjects will be taking half a Carvedilol per day at first week and one Carvedilol per day from second week. At the same time,the subjects will be taking one Entecavir tablet per day for 96 weeks.
  Arms: Entecavir/Carvedilol
Drug: Entecavir+Carvedilol+ Fuzheng Huayu — The subjects will be taking half a Carvedilol tablet per day at first week and one Carvedilol tablets per day from second week. At the same time,the subjects will be taking one Entecavir tablet per day and 4 Fuzheng Huayu tablets three times a day for 96 weeks.
  Arms: Entecavir/Carvedilol/ Fuzheng Huayu

SUMMARY:
Portal hypertension is a common pathology in chronic liver disease, particularly in liver cirrhosis. Hepatitis B Virus (HBV) is one of most etiologies of liver cirrhosis in China. The basic reason for portal hypertension in HBV is the largely deposition of hepatic extracellular matrixes which causes high pressure in liver vessels. One of the most common symptoms of cirrhotic portal hypertension is gastroesophageal varices.The effective inhibition of HBV can partially stop or reverse liver fibrosis in patients with chronic Hepatitis and liver cirrhosis due to HBV and the anti-fibrotic strategy focusing on the regulation of hepatic extracellular matrix may have a great benefit. Therefore, antivirals therapy is also a basic treatment for low-grade cirrhotic portal hypertension. Fuzheng Huayu has been found to enhance the degradation of collagens in fibrotic liver and have a good action against liver fibrosis in patients with chronic hepatitis B. However, there are no high quality clinical evidences which can demonstrate if the combination of anti-viral and anti-fibrotic therapy can relieve the pressure of liver vessels and decline incidence rate and bleeding rate of gastroesophageal varices.

DETAILED DESCRIPTION:
The primary objective of this study is to establish the safety and efficacy of the combination of Entecavir and Fuzheng Huayu for reverse rate of gastroesophageal varices in patients with Moderate and Severe cirrhotic portal hypertension due to hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

* More than 6 months history of serum positive HBsAg
* Abdominal ultrasonogram or CT scan or liver-biopsy specimen indicates liver cirrhosis
* Age 18-65
* Child-Pugh<7 (Stage A)
* Without portal hypertension（Endoscopy indicates no signs of gastroesophageal varices.）
* Moderate and Severe of portal hypertension（Endoscopy indicates signs of gastroesophageal varices that is line shape without red wales or spots and less than 0.3cm of diameter.）
* The patient or the patient's guardian agrees to participate the random controlled trial and sign the Informed Consent Form.

Exclusion Criteria:

* Primary Lamivudine, Adefovir dipivoxil and Entecavir resistance
* Decompensated cirrhosis、The Child-Pugh score≥7
* Low-grade Cirrhotic Portal Hypertension.
* Severe grade of portal hypertension（Endoscopy indicates signs of gastroesophageal varices that is catenulate/nodular shape with or without red wales or spots and more than 1.0cm of diameter.）
* Decompensated liver cirrhosis Liver cancer
* Liver histology conforming to other chronic liver diseases, such as moderate or severe non-alcoholic fatty liver disease(more than 1/3 steatosis in liver ), chronic hepatitis C, chronic hepatitis D, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, inherited metabolic liver disease, drug or toxic induced liver injury, parasitic infections, alcoholic liver disease.
* Have psychiatric history or uncontrollable epilepsy patient.
* Uncontrollable diabetic patient
* History of hemoglobin disease (such as alpha- or beta-thalassemia, sickle cell disease, spherocytosis) or patients with toxic or autoimmune hemolytic anemia.
* Severe background disease like chronic respiratory failure, circulatory failure, kidney failure etc.
* In situ organ transplantation (such as liver, kidney, lung and heart) or bone marrow transplantation and stem cell transplantation.
* Immunocompromised patients: such as HIV infection or take immunosuppressor or glucocorticoid (such as cyclosporin, azathioprine, adrenocortical hormone) within 3 months or chemotherapy drugs (such as cyclophosphamide, ammonia and cancer chemotherapy) and radioactive therapy.
* Gestation or lactation period women and women who plan to get pregnant during the study period.
* Patient who are allergy to the experimental drug.
* Using history of anti-viral or anti-fibrosis drug within 6 months.
* Patients who are participating other trials.
* Other situation where PI thinks the patient should be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical events: Variceal hemorrhage, Ascites, Encephalopathy, etc | 96 weeks
Grading varices | 96 weeks
Incidence of liver cancer | 96 weeks
Noninvasive portal hypertension index | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: CHENGHAI LIU, PHD,MD, Principal Investigator — ShuGuang Hospital
Locations (3):
- China (3):
  - Ruijin Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided